CLINICAL TRIAL: NCT04673149
Title: Multicenter, Randomized, Combined Phase I Dose-escalation and Phase IIa Double-blind, Placebo-controlled Study of the Safety, Tolerability, and Immunogenicity of GLS-5310 DNA Vaccine, Administered Intradermally Against SARS-CoV-2 in Healthy Adults
Brief Title: GLS-5310 Vaccine for the Prevention of SARS-CoV-2 (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CoV2-001
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV-2
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — GLS-5310 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GLS-5310 0.6mg [Group 1a] (Experimental): 0.6mg of GLS-5310 will be intradermally administered on Day 0 and Week 8.
  Interventions: Biological: GLS-5310
- GLS-5310 1.2mg [Group 1b] (Experimental): 1.2mg of GLS-5310 will be intradermally administered on Day 0 and Week 8.
  Interventions: Biological: GLS-5310
- GLS-5310 1.2mg [Group 1c] (Experimental): 1.2mg of GLS-5310 will be intradermally administered on Day 0 and Week 12.
  Interventions: Biological: GLS-5310
- Placebo [Group 2a] (Placebo Comparator): Placebo will be intradermally administered on Day 0 and Week 8 (or Week 12).
  Interventions: Biological: Placebo
- GLS-5310 1.2mg [Group 2b] (Experimental): 1.2mg of GLS-5310 will be intradermally administered on Day 0 and Week 8 (or Week 12).
  Interventions: Biological: GLS-5310

INTERVENTIONS:
Biological: GLS-5310 — GLS-5310 DNA plasmid vaccine
  Arms: GLS-5310 0.6mg [Group 1a]; GLS-5310 1.2mg [Group 1b]; GLS-5310 1.2mg [Group 1c]; GLS-5310 1.2mg [Group 2b]
Biological: Placebo — Placebo
  Arms: Placebo [Group 2a]

SUMMARY:
This clinical trial will evaluate the safety, tolerability and immunogenicity of GLS-5310 DNA vaccine against SARS-CoV-2(COVID-19) in healthy volunteers.

DETAILED DESCRIPTION:
This Phase I / IIa study will assess the safety, tolerability, and immunogenicity of GLS-5310 DNA vaccine.

The Phase I portion of this study is an open-label, dose escalation study to assess two dose levels of GLS-5310 DNA vaccine (0.6 and 1.2 mg) as part of two vaccination regimens (0-8 weeks and 0-12 weeks).

The Phase IIa portion of this study is designed as a randomized, double-blind, placebo-controlled study with only a single active study drug arm. Subjects will be randomized to receive either placebo or GLS-5310 vaccine in a 1:2 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 to 85 years of age (Phase I will be restricted to an upper age limit of 50 years of age)
2. Able to provide informed consent
3. Able and willing to comply with study procedures
4. For women of childbearing potential, able and willing to use an approved form of pregnancy prevention through to 4 weeks post boost vaccination

Exclusion Criteria:

1. Current or planned pregnancy through to 4 weeks post-boost vaccination for women of childbearing potential
2. Currently breastfeeding
3. Current or past participation in a coronavirus (MERS-CoV, SARS-CoV-2) vaccine study
4. Administration of an investigational agent within 6 months of the 1st dose
5. Administration of a vaccine within 4 weeks prior to the 1st dose
6. Administration of immune globulin within 16 weeks of enrollment
7. Administration of an anti-TNFα inhibitor such as infliximab, adalimumab, etanercept, or anti-CD20 monoclonal antibody rituximab within 24 weeks prior to enrollment
8. Current daily treatment of systemic corticosteroids of 20 mg of prednisone or greater, dexamethasone of 3 mg or greater; or the equivalent dose of other systemic corticosteroids
9. Administration of any Immunosuppressive Drug or Immunomodulator within 3 months of the first dose
10. History of bone marrow transplantation
11. Current or planned chemotherapy treatment for hematologic or solid tumor during study period or treatment during the 5 years prior to enrollment
12. Respiratory disease (ex. Asthma, Chronic obstructive lung disease)
13. Cardiovascular disease (ex. myocardial ischemia, congestive heart failure, cardiomyopathy, clinically significant arrhythmia)
14. Hypertension (Systolic pressure >150mmHg or Diastolic pressure >95mmHg)
15. Confirmed Diabetes
16. Severe allergic reaction or anaphylactic reaction after vaccination in the past
17. Immunosuppresion including immunodeficiency disease or family history
18. Positive of serum test at screening (Hepatitis B, Hepatitis A, HIV, Hepatitis C)
19. Baseline screening lab(s) with Non Clinical Significant abnormality
20. Serious adverse reaction to a drug containing Investigational Product (GLS-5310) or other ingredients of the same categories or to a vaccine or antibiotic, nonsteroidal anti-inflammatory disease control, etc. or an allergic history
21. History of hypersensitivity to vaccination such as Guillain-Barre syndrome
22. History of PCR-confirmed infection with SARS-CoV-2 at screening
23. Subjects who have been contact with COVID-19 infections in the past prior to administration, have been classified as COVID-19 confirmed patients, medical patients or patients with symptoms or have been identified with SARS and MERS infection history in the past
24. 37.5 degrees, cough, difficulty breathing, chills, muscle aches, headache, sore throat, loss of smell, or loss of taste within 72 hours prior to administration
25. Healthcare workers participating in the medical examination of patients infected with COVID-19
26. Not willing to allow storage and future use of samples for SARS-CoV-2 related research
27. Prisoner or subjects who are compulsorily detained for treatment of a psychiatric illness
28. Any illness or condition that, in the opinion of the investigator, may affect the safety of the subject or the evaluation of a study endpoint

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GLS-5310 0.6mg [Group 1a] | GLS-5310 1.2mg [Group 1b] | GLS-5310 1.2mg [Group 1c] | Placebo [Group 2a] | GLS-5310 1.2mg [Group 2b]
Started | 15 | 15 | 15 | 42 | 84
Completed | 15 | 15 | 15 | 26 | 77
Not Completed | 0 | 0 | 0 | 16 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLS-5310 0.6mg [Group 1a] | GLS-5310 1.2mg [Group 1b] | GLS-5310 1.2mg [Group 1c] | Placebo [Group 2a] | GLS-5310 1.2mg [Group 2b] | Total
Number analyzed (Participants) | 15 | 15 | 15 | 42 | 84 | 171
Age, Customized [Count of Participants; unit: Participants]
  Age 19-66 | 15 | 15 | 15 | 42 | 80 | 167
  Age >66-85 | 0 | 0 | 0 | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 14 | 31 | 64 | 127
  Male | 6 | 6 | 1 | 11 | 20 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 15 | 15 | 42 | 84 | 171
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events
Time Frame: Through 48 weeks post vaccination
Measure: Number; unit: serious adverse events
Arm/Group | GLS-5310 0.6mg [Group 1a] | GLS-5310 1.2mg [Group 1b] | GLS-5310 1.2mg [Group 1c] | Placebo [Group 2a] | GLS-5310 1.2mg [Group 2b]
Number analyzed (Participants) | 15 | 15 | 15 | 42 | 84
serious adverse events | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Positive T Cell Responses Induced by GLS-5310
Time Frame: Post vaccination Visit 4 (4 weeks after week 8 or week 12 vaccination)
Measure: Count of Participants; unit: Participants
Arm/Group | GLS-5310 0.6mg [Group 1a] | GLS-5310 1.2mg [Group 1b] | GLS-5310 1.2mg [Group 1c] | Placebo [Group 2a] | GLS-5310 1.2mg [Group 2b]
Number analyzed (Participants) | 15 | 15 | 15 | 38 | 75
Participants | 14 | 12 | 14 | 14 | 24

3. Secondary Outcome: Number of Participants With Positive Neutralizing Antibody Responses Induced by GLS-5310
Time Frame: Post vaccination Visit 4 (4 weeks after week 8 or week 12 vaccination)
Measure: Count of Participants; unit: Participants
Arm/Group | GLS-5310 0.6mg [Group 1a] | GLS-5310 1.2mg [Group 1b] | GLS-5310 1.2mg [Group 1c] | Placebo [Group 2a] | GLS-5310 1.2mg [Group 2b]
Number analyzed (Participants) | 15 | 15 | 15 | 38 | 75
Participants | 4 | 5 | 6 | 2 | 7

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from Week 0 through Week 48.
Description: Adverse events were graded according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials guidelines that were issued by the Food and Drug Administration in September 2007.
Arm/Group | GLS-5310 0.6mg [Group 1a] | GLS-5310 1.2mg [Group 1b] | GLS-5310 1.2mg [Group 1c] | Placebo [Group 2a] | GLS-5310 1.2mg [Group 2b]
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/44 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/44 | 0/82
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 15/15 | 33/44 | 82/82
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLS-5310 0.6mg [Group 1a] (N=15) | GLS-5310 1.2mg [Group 1b] (N=15) | GLS-5310 1.2mg [Group 1c] (N=15) | Placebo [Group 2a] (N=44) | GLS-5310 1.2mg [Group 2b] (N=82)
Injection site erythyma (General disorders) | 9 (9) | 13 (13) | 14 (14) | 15 (15) | 55 (55)
Injection site pruritus (General disorders) | 9 (9) | 11 (11) | 10 (10) | 5 (5) | 33 (33)
Injection site edema (General disorders) | 4 (4) | 10 (10) | 7 (7) | 5 (5) | 28 (28)
Injection site pain (General disorders) | 1 (1) | 2 (2) | 3 (3) | 8 (8) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT04673149/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT04673149/SAP_001.pdf